CLINICAL TRIAL: NCT04192669
Title: Study of Heart Rate Variability as a Clinical Marker in a Population of Anxio-depressive Patients
Brief Title: Heart Rate Variability as a Clinical Marker in a Population of Anxio-depressive Patients
Status: Completed | Type: Observational
Sponsor: Tatiana Besse-Hammer (Other)
Responsible Party: Sponsor-Investigator, Tatiana Besse-Hammer, Head of clinical research unit, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-PSY-BRUHRV
Record Dates: First submitted 2019-12-05; First posted 2019-12-10 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Anxio Depressive Disorder
MeSH Terms: interventions — Heart Rate Determination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anxio-depressive patients: Patients with a depressive or anxious disorder going to the Psychiatry Department of the CHU Brugmann Hospital.
  Interventions: Device: Heart rate monitoring

INTERVENTIONS:
Device: Heart rate monitoring — The heart rate will be recorded and calculated by a heart rate monitor (Polar H10, Finland) located on the chest. The recording is done over a period of 5 minutes, the patient being in a sitting position, without any particular stimulus, in a quiet room. The recording is transferred via the HRV Logger application. Any ectopic beats and artifacts are automatically identified and replaced by values interpolated by the investigator, if necessary. The Kubios HRV Premium Software is used for all calculations.

SUMMARY:
The heart rate (HR) is regulated by the autonomic nervous system (ANS) and results from a balance between the sympathetic nervous system (SNS) that accelerates the heart rate and the parasympathetic nervous system that slows the HR via the vagus nerve.

Low HRV is linked to poor emotional and cognitive regulation. Values for HRV are generally lower in depressed patients.

The aim of this study is to determine how HRV could be a clinical marker that can be used in routine psychiatry practice in patients with anxio-depressive disorders, to determine the severity of symptoms and the degree of response to treatment.

ELIGIBILITY:
Inclusion Criteria:

- Patients of the CHU Brugmann Hospital with an anxious or depressive disorder

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the Psychiatry Department of the CHU Brugmann Hospital with an anxious or depressive disorder.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
Beck depression inventory (BDI) | Baseline (day of inclusion of the patient in the study).
  Multiple choice (4 choices) questionnaire with 21 items. The end score can vary between 0 and 63. Score interpretation: 1-10: These ups and downs are considered normal. 11-16 Mild mood disturbance. 17-20 Borderline clinical depression. 21-30 Moderate depression. 31-40 : Severe depression. Over 40 :Extreme depression.
Beck depression inventory (BDI) | Measured only once at one visit taking place minimum 3 months and maximum 6 months after baseline
  Multiple choice (4 choices) questionnaire with 21 items. The end score can vary between 0 and 63. Score interpretation: 1-10: These ups and downs are considered normal. 11-16 Mild mood disturbance. 17-20 Borderline clinical depression. 21-30 Moderate depression. 31-40 : Severe depression. Over 40 :Extreme depression.
State trait Anxiety inventory (STAI) | Baseline (day of inclusion of the patient in the study).
  The State-Trait Anxiety Inventory (STAI) is a psychological inventory based on a 4-point Likert scale and consists of 40 questions on a self-report basis. Scores range from 20 to 80, with higher scores correlating with greater anxiety.
State trait Anxiety inventory (STAI) | Measured only once at one visit taking place minimum 3 months and maximum 6 months after baseline
  The State-Trait Anxiety Inventory (STAI) is a psychological inventory based on a 4-point Likert scale and consists of 40 questions on a self-report basis. Scores range from 20 to 80, with higher scores correlating with greater anxiety.
Maslach Burnout inventory (MBI) | Baseline (day of inclusion of the patient in the study).
  The Maslach Burnout Inventory (MBI) is an introspective psychological inventory consisting of 22 items pertaining to occupational burnout. All MBI items are scored using a 7 level frequency scale from "never" to "daily." Initial development had 3 components: emotional exhaustion (9 items), depersonalization (5 items) and personal achievement (8 items). Each scale measures its own unique dimension of burnout. Scales should not be combined to form a single burnout scale.
Maslach Burnout inventory (MBI) | Measured only once at one visit taking place minimum 3 months and maximum 6 months after baseline
  The Maslach Burnout Inventory (MBI) is an introspective psychological inventory consisting of 22 items pertaining to occupational burnout. All MBI items are scored using a 7 level frequency scale from "never" to "daily." Initial development had 3 components: emotional exhaustion (9 items), depersonalization (5 items) and personal achievement (8 items). Each scale measures its own unique dimension of burnout. Scales should not be combined to form a single burnout scale.
Root mean square of successive differences (RMSSD) | Baseline (day of inclusion of the patient in the study).
  The Root Mean Square of the Successive Differences (RMSSD) is one of a few time-domain tools used to assess heart rate variability, the successive differences being neighboring RR intervals. It reflects the activity of the parasympathetic nervous system.
Root mean square of successive differences (RMSSD) | Measured only once at one visit taking place minimum 3 months and maximum 6 months after baseline
  The Root Mean Square of the Successive Differences (RMSSD) is one of a few time-domain tools used to assess heart rate variability, the successive differences being neighboring RR intervals. It reflects the activity of the parasympathetic nervous system.
High frequency percentage in the spectral analysis of the heart RR interval | Baseline (day of inclusion of the patient in the study).
  Spectral analysis of the RR interval is an indirect, noninvasive measurement tool of heart rate variability. High-frequency RR signals (0.15 to 0.4 Hz) reflect a parasympathetic activity and thus an influence of the vagal nerve on the heart. A high frequency heart variability is associated with a better perception of emotions and with pro-social behaviors.
High frequency percentage in the spectral analysis of the heart RR interval | Measured only once at one visit taking place minimum 3 months and maximum 6 months after baseline
  Spectral analysis of the RR interval is an indirect, noninvasive measurement tool of heart rate variability. High-frequency RR signals (0.15 to 0.4 Hz) reflect a parasympathetic activity and thus an influence of the vagal nerve on the heart. A high frequency heart variability is associated with a better perception of emotions and with pro-social behaviors.

SECONDARY OUTCOMES:
Toronto Alexithymia scale (TAS 20) | Baseline (day of inclusion of the patient in the study).
  The TAS is a 20-item instrument that is one of the most commonly used measures of alexithymia. Alexithymia refers to people who have trouble identifying and describing emotions and who tend to minimise emotional experience and focus attention externally. The TAS-20 uses cutoff scoring: equal to or less than 51 = non-alexithymia, equal to or greater than 61 = alexithymia. Scores of 52 to 60 = possible alexithymia.
Toronto Alexithymia scale (TAS 20) | Measured only once at one visit taking place minimum 3 months and maximum 6 months after baseline
  The TAS is a 20-item instrument that is one of the most commonly used measures of alexithymia. Alexithymia refers to people who have trouble identifying and describing emotions and who tend to minimise emotional experience and focus attention externally. The TAS-20 uses cutoff scoring: equal to or less than 51 = non-alexithymia, equal to or greater than 61 = alexithymia. Scores of 52 to 60 = possible alexithymia.
Difficulties in Emotion Regulation Scale (DERS-18) | Baseline (day of inclusion of the patient in the study).
  The Difficulties in Emotion Regulation Scale is a self-report measure that evaluates individuals' levels of difficulties in regulating emotions.Higher scores indicate more difficulty in emotion regulation.
Difficulties in Emotion Regulation Scale (DERS-18) | Measured only once at one visit taking place minimum 3 months and maximum 6 months after baseline
  The Difficulties in Emotion Regulation Scale is a self-report measure that evaluates individuals' levels of difficulties in regulating emotions.Higher scores indicate more difficulty in emotion regulation.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Cole, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No